CLINICAL TRIAL: NCT04742621
Title: Liver Transplantation for Unresectable Liver Limited Colorectal Metastases
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 20-04021768
Record Dates: First submitted 2021-01-22; First posted 2021-02-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Unresectable Liver-limited Colorectal Metastases
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Liver transplant — Eligibility for liver transplantation will be limited to patients with histologically confirmed metastatic colorectal adenocarcinoma who have achieved stability of liver metastasis on chemotherapy for at least 6 months prior to transplantation. All patients who undergo liver transplantation will start immunosuppressive therapy per protocol. Patients who undergo a successful liver transplant will not receive adjuvant therapy.

SUMMARY:
This is a single-arm, single institution pilot registry of liver transplantation in patients with unresectable colorectal liver-only metastases at Weill Cornell Medical College. Patients with liver predominant colorectal liver metastases will be screened based on eligibility criteria in a specified clinical hepatobiliary and colorectal liver metastasis tumor board consisting of the principal and co-investigators, representing medical oncology, transplant surgery, radiology, and pathology. The registry aims to track basic demographic data as well as referral patterns, in addition to specific oncologic data such as tumor burden, extent of disease, extent of disease on explant, recurrence rates, patterns of recurrence and survival rates.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the colon or rectum
2. No evidence of extrahepatic metastases or local recurrence based on PET/CT and colonoscopy
3. No signs of extrahepatic metastases or local recurrence according to PET/CT 4 weeks prior to consideration of transplant
4. Age 18-65 years old
5. Good performance status with ECOG 0-1
6. Stability or regression of liver metastasis for at least 6 months
7. Minimum of 1 year between diagnosis of colon cancer and liver transplant and 6 months from primary tumor resection and liver transplant
8. Minimum of 6 months chemotherapy
9. CEA < 200 ug/L 3 months prior to transplant
10. Adequate organ and marrow function with Hb > 10 g/dL, ANC > 1000/uL, platelets > 100,000/uL, bilirubin < 2x ULN, AST/ALT < 5x ULN, Creatinine < 1.25 x ULN, Albumin above LLN

Exclusion Criteria:

1. Evidence of extrahepatic disease or local recurrence
2. Previous resection of lung metastases
3. MSI-H/dMMR or BRAF mutation
4. Any other medical or co-morbid condition that would preclude liver transplantation, as determined by the transplant team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver predominant colorectal liver metastases will be screened based on eligibility criteria in a specified clinical hepatobiliary and colorectal liver metastasis tumor board. If deemed acceptable candidates for liver transplantation, they will then undergo transplant evaluation as per Weill Cornell Medical College Liver Transplant clinical protocols.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2034-07-27 (Estimated); Study Completion 2035-07-27 (Estimated)

PRIMARY OUTCOMES:
To develop a registry of liver transplantation in patients with liver limited metastatic colorectal cancer at Weill Cornell Medical College / New York-Presbyterian Hospital (WCMC / NYPH) | 25 years

SECONDARY OUTCOMES:
To determine disease-free survival (DFS) in patients that receive a liver transplant for metastatic colorectal cancer at Weill Cornell Medical College / New York-Presbyterian Hospital | 25 years
To determine overall survival (OS) in patients that receive a liver transplant for metastatic colorectal cancer at Weill Cornell Medical College / New York-Presbyterian Hospital | 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Samstein, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No